CLINICAL TRIAL: NCT07267338
Title: Pembrolizumab Combined With MRG-003 as Neoadjuvant Treatment of EBV- Associated Locoregionally Advanced Nasopharyngeal Carcinoma: A Single-arm, Single-center, Prospective Phase II Trial
Brief Title: Pembrolizumab + MRGOO3 as Neoadjuvant in NPC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISP102452
Record Dates: First submitted 2025-07-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: NPC; Locoregionally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Participants will receive 3 cycles of neoadjuvant Pembrolizumab 200 mg IV every 3 weeks (Q3W) combined MRG003 2.0mg/kg IV Q3W followed by standard CCRT and adjuvant treatment of Pembrolizumab 200 mg IV Q3W up to 14 cycles.
  Interventions: Drug: Pembrolizumab & MRG003

INTERVENTIONS:
Drug: Pembrolizumab & MRG003 — After a screening phase of up to 28 days, each subject will be assigned to receive treatment until disease progression is confirmed, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, or until subjects has received up to 3 cycles pembrolizumab + MRG003, followed Standard concurrent chemoradiotherapy (CCRT), followed up to 14 cycles pembrolizumab.

SUMMARY:
The goal of this clinical trial is to evaluate efficacy and safety of neoadjuvant of the anti PD1 agent Pembrolizumab combined with MRG003 and adjuvant treatment of Pembrolizumab in patients with Epstein-Barr virus (EBV) - associated locoregionally advanced nasopharyngeal carcinoma.

The expected sample size is 35 patients.

Participants will receive 3 cycles of neoadjuvant pembrolizumab 200mg Q3W plus MRG003 2.3mg/kg Q3W followed by the standard concurrent chemoradiotherapy. Then participants will receive 14 cycles of adjuvant Pembrolizumab 200 mg Q3W after the standard concurrent chemoradiotherapy.

The estimated average length of treatment per patients is 1 year.

DETAILED DESCRIPTION:
This is a prospective, single-group, open-label, phase II trial to evaluate the efficacy and safety of 3 cycles of neoadjuvant pembrolizumab and MRG003 followed by concurrent CCRT and 14 cycles of adjuvant pembrolizumab in EBV-associated locoregionally advanced nasopharyngeal carcinoma patients.

The primary objective is to evaluate the Clinical Complete Response (cCR) rate of neoadjuvant pembrolizumab+MRG003 in EBV-associated locoregionally advanced nasopharyngeal carcinoma. The CT/MRI head and neck, chest, upper abdomen for cCR assessment will be performed on week 9±7 days between neoadjuvant therapy and pre CCRT.

Each subject will participate in the trial from the time the subject signs the informed consent form (ICF) through the final protocol-specified contact.

After a screening phase of up to 28 days, each subject will be assigned to receive treatment until disease progression is confirmed, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, or until subjects has received up to 3 cycles pembrolizumab + MRG003, followed Standard concurrent chemoradiotherapy (CCRT), followed up to 14 cycles pembrolizumab (approximately 1 year).

After the end of treatment, each subject will be followed for the occurrence of adverse events.

Subjects who discontinue for reasons other than disease progression will have post-treatment follow-up for disease status until disease progression is confirmed by the site per RECIST 1.1, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone for overall survival until death, withdrawal of consent or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of stage III-IVa (Exclude T3N0) nasopharyngeal carcinoma (NPC) will be enrolled in this study.
2. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
3. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
4. Archival tumor tissue sample or newly obtained [core or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slide. Newly obtained biopsies are preferred to archived tissue.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
6. Epsitein-Barr virus-encoded RNA(EBER) positive.
7. Epidermal Growth Factor Receptor (EGFR) positive.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
10. Have adequate organ function. Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

1. Presence of any distant metastasis.
2. Has received prior therapy with EGFR target therapy, or an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to [allocation].
4. Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
5. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
6. Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤6, and PSA <10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab, MRG003 and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. History of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as detectable HCV RNA [qualitative]) infection.

    Note: Testing for Hepatitis B or C is not required unless mandated by local health authority.
15. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by local health authority
16. Has not adequately recovered from major surgery or has ongoing surgical complications.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has had an allogenic tissue/solid organ transplant.
21. History of HIV infection. HIV testing is not required unless mandated by local health authority.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Complete Response (cCR) rate | cCR assessment will be performed on week 9±7 days between neoadjuvant therapy and pre CCRT
  clinical complete response (cCR) rate to neoadjuvant treatment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | To assess the objective response rate of Neoadjuvant therapy of Pembrolizumab in combination with MRG003 at maximum of 9 weeks (up to 3 cycles)
  ORR, defined as the proportion of participants who have achieved a confirmed complete response (CR), or partial response (PR), which is assessed according to RECIST 1.1 criterial.
Event-Free Survival (EFS) | Defined as the time from date of treatment to the date of first documented disease progression that precluded definitive surgery, local or distant recurrence, occurrence of a second primary cancer or death from any cause, up to 36 months
  To evaluate neoadjuvant therapy of Pembrolizumab in combination with MRG003 and adjuvant therapy of Pembrolizumab with respect to event-free survival (EFS).
Overall Survival (OS) | OS, defined as the time from the date of treatment to the date of death due to any cause, up to 60 months
  To evaluate neoadjuvant therapy of Pembrolizumab in combination with MRG003 and adjuvant therapy of Pembrolizumab with respect to overall survival (OS).

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Xiehe Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No